CLINICAL TRIAL: NCT06823401
Title: IMMUNOBLOOD: Perspective Study for the Evaluation of Anti-Inhibitory Checkpoint Antibody Development in Patients Undergoing Immunotherapy
Brief Title: Study Investigating Anti-drug Antibodies in NSCLC Patients Exposed to Checkpoint Inhibitors (IMB)
Acronym: IMB
Status: Recruiting | Type: Observational
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Other Study IDs: IMMUNOBLOOD; RS1466/21(2477) (Other: Fondazionefort)
Record Dates: First submitted 2025-01-13; First posted 2025-02-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: NSCLC
Keywords: immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Plasma levels of anti-drug antibodies will be analyzed prior trial therapy and prior each next cycle until disease progression.
  Blood sample (6 ml) will be collected by enrolled patients and spinned at 1500 rpm (within 2/3 24 hours the withdrawal) at Regina Elena National Cancer Institute (IRE).
  In particular, plasma levels of anti-drug antibodies will be assessed by using enzyme immunoassay (ELISA). The method employs the principle of competitive ELISA, allowing quantification of anti-drug antibodies (expressed in µg/ml), according to an internal standard curve.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-small cell lung cancer (NSCLC) is one of the leading causes of death in Western countries. Today, a new frontier in the fight against cancer is immunotherapy, a treatment that aims to "awaken" the patient's immune system to help it recognize and attack cancer cells.

Among the various approaches, there is significant focus on therapies that activate T lymphocytes, a type of immune cell, encouraging them to react against the tumor. These treatments have led to important progress and represent a hope for the future.

DETAILED DESCRIPTION:
Prospective study aimed at evaluating the development of anti-drug antibodies in patients with NSCLC treated with immune checkpoint inhibitors, either as monotherapy or in combination, and the correlation between the presence of anti-drug antibodies, treatment efficacy, and the occurrence of adverse drug reactions.

Primary objective:

To assess whether patients treated with checkpoint inhibitors as single agent or in combination with other checkpoint inhibitors or chemotherapy develop anti-drug antibodies during the course of treatment Secondary objective: To assess whether development of anti-drug antibodies is associated with response, duration of response, PFS, OS, toxicity For each eligible patient, a blood sample (6 ml) will be collected before the start of therapy and before each treatment cycle until disease progression or the completion of the planned cycles. The tests and procedures the patient will undergo are all considered routine and part of standard medical care, so they do not entail any additional risks associated with participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC
* Possibility to obtain blood samples
* Patient candidate, in any therapy line, for a therapy with any checkpoint inhibitor including single agent pembrolizumab, single agent atezolizumab, single agent nivolumab, single agent durvalumab or combination of nivolumab and ipilimumab
* Performance status 0-2 (ECOG)
* Patient compliance to trial procedures
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* No possibility to obtain blood samples
* Previous therapy with any checkpoint inhibitor
* Patient candidate for a therapy with a checkpoint inhibitor in combination with chemotherapy or any other non-checkpoint inhibitors
* Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include NSCLC patients candidate, in any therapy line, for a therapy with any checkpoint inhibitor including single agent pembrolizumab, single agent atezolizumab, single agent nivolumab, single agent durvalumab or combination of nivolumab and ipilimumab
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Anti-Checkpoint Inhibitor Antibodies in Plasma of Participants Receiving Treatment | From the start of treatment until the first documented progression, completion of treatment cycles, or death from any cause, whichever occurs first, assessed from the start of treatment up to 12 months.
  Detection of anti-checkpoint inhibitors antibodies in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Federico FC Cappuzzo, PI, Principal Investigator — IRCCS Ist. Naz. Tum. Regina Elena
Locations (1):
- Istituto Tumori Regina Elena, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided